CLINICAL TRIAL: NCT00307203
Title: Nicotine and Smoking Cessation in Schizophrenia
Brief Title: Safety and Effectiveness of Sustained Release Bupropion in Treating Individuals With Schizophrenia Who Smoke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Ivan Montoya, NIDA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23DA000510 (NIH); DPMC
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-09

CONDITIONS: Tobacco-Use Disorder; Schizophrenia; Psychotic Disorders
Keywords: Bupropion; Zyban; Wellbutrin; Smoking cessation; Schizophrenia; Schizoaffective disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Psychotic Disorders; Smoking Cessation | interventions — Bupropion; Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Experiment group received 300 mgs of bupropion, in addition to weekly CBT and nicotine replacement therapy
  Interventions: Drug: bupropion SR; Behavioral: Cognitive Behavioral Group Therapy; Drug: nicotine replacement therapy
- II (Placebo Comparator): Placebo group received placebo, in addition to weekly CBT and nicotine replacement therapy
  Interventions: Behavioral: Cognitive Behavioral Group Therapy; Drug: nicotine replacement therapy

INTERVENTIONS:
Drug: bupropion SR — Participants were randomly assigned to receive bupropion SR 150 mg or placebo, once daily for 7 days, then twice daily for 11 weeks.
  Other Names: Zyban, Wellbutrin
  Arms: I
Behavioral: Cognitive Behavioral Group Therapy — Participants attended a 12-session, 1-hour, weekly smoking cessation group program with 3 to 7 participants led by a psychologist with tobacco treatment specialist training. Subjects set a quit date, and nicotine patches (Habitrol) and nicotine polacrilex gum (Nicorette) were initiated in the fourth week.
  Other Names: CBT
Drug: nicotine replacement therapy — Nicotine patch was dosed at 21 mg/d for 4 weeks, 14 mg/d for 2 weeks, and 7 mg/d for 2 weeks, then discontinued. Nicotine gum (2 mg) was distributed for use as needed for craving up to 18 mg/d.
  Other Names: nicotine patch; nicotine gum

SUMMARY:
Many individuals with schizophrenia smoke cigarettes. Individuals in the schizophrenic population often find it difficult to quit smoking. The purpose of this trial is to determine the safety and effectiveness of bupropion in treating individuals with schizophrenia who smoke.

DETAILED DESCRIPTION:
Schizophrenia affects 1 % of the population. Among individuals with schizophrenia, between 74 and 92 % smoke cigarettes regularly. Heavy smoking represents a significant and neglected public health problem for people with schizophrenia; smoking cessation treatment is often overlooked as part of the psychiatric care for such individuals.

The most effective treatment for smoking cessation described to date is sustained release (SR) bupropion. Past research suggests that SR bupropion may be especially effective in individuals with depressive symptoms, including individuals with schizophrenia. The purpose of this trial is to evaluate the safety and efficacy of SR bupropion, when combined with cognitive behavioral therapy (CBT), in individuals with schizophrenia.

This trial will last 12 weeks. Participants will be randomly assigned to receive SR bupropion or placebo. All participants will receive weekly CBT. Participants will be followed for 3 months following completion of the 12-week treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia or schizoaffective disorder
* Receiving a stable dose of antipsychotic medication for at least 1 month prior to study entry
* Smokes at least 10 cigarettes per day
* Wishes to stop smoking
* Attended last three scheduled clinic visits, prior to study entry

Exclusion Criteria:

* Significant medical or neurologic illness
* History of severe head injury with loss of consciousness
* Treated with monoamine oxidase inhibitors or carbamazepine in the 14 days prior to study entry
* Taking clozapine at doses greater than 500 mg/d without an anticonvulsant
* Currently undergoing an acute exacerbation of psychotic symptoms
* Current or history of bulimia or anorexia
* Current excessive water intake
* Recent history of mania
* Known allergy or hypersensitivity to bupropion
* Current substance abuse other than tobacco, nicotine replacement treatment, or smokeless tobacco
* Currently receiving treatment with bupropion
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1998-08; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
seven-day point prevalence of smoking reduction, defined as 50 % reduction in serum cotinine levels compared to baseline | end of treatment

SECONDARY OUTCOMES:
continuous smoking reduction (50 % reduction in weekly expired air carbon monoxide (CO) measurements compared to baseline and self report) | end of treatment
continuous tobacco abstinence (weekly expired CO measurements less than 9 ppm and self report) | end of treatment
psychotic symptoms | continuous and end of treatment
negative side effects | continuous
negative and depressive symptoms compared to baseline at the end of the 3-month treatment and 3-month follow-up phases | continuous and end of treatment
measures of attention and memory while attempting to quit smoking | end of treatment
health-related quality at the end of the 3-month treatment and 3-month follow-up phases | continuous and end of treatment
weight gain at the end of the 3-month treatment and 3-month follow-up phases | continuous and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: A Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Result] Evins AE, Cather C, Culhane MA, Birnbaum A, Horowitz J, Hsieh E, Freudenreich O, Henderson DC, Schoenfeld DA, Rigotti NA, Goff DC. A 12-week double-blind, placebo-controlled study of bupropion sr added to high-dose dual nicotine replacement therapy for smoking cessation or reduction in schizophrenia. J Clin Psychopharmacol. 2007 Aug;27(4):380-6. doi: 10.1097/01.jcp.0b013e3180ca86fa. PMID 17632223
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961